CLINICAL TRIAL: NCT00651417
Title: A Phase II, Pilot, Randomized, Double-blind Study Comparing the Effectiveness Organic Germanium to Placebo in Decreasing the Severity of Fatigue in Patients Undergoing Radiation Therapy for Prostae and Bbreast Cancers
Brief Title: Use of Organic Germanium or Placebo for the Prevention of Radiation Induced Fatigue
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arizona Oncology Services (Other)
Responsible Party: Emily Grade,M.D., Principal Investigator, Arizona Oncology Serivces Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Germanium
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Localized Breast Cancer; Localized Prostate Cancer; Patients Receiving External Beam Radiotherapy
Keywords: Organic germanium; fatigue; radiation therapy; breast cancer; prostate cancer
MeSH Terms: conditions — Fatigue; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Organic Germanium tablets 5 times a day
  Interventions: Dietary Supplement: Organic Germanium
- 2 (Placebo Comparator): Placebo tablets 3 -5 times per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Organic Germanium — Oral organic Germaium tablets on the tongue 3 to 5 times per day as tolerated
  Other Names: Allergy Research Group supplies the organic Germanium
  Arms: 1
Dietary Supplement: Placebo — Placebo tablets orally 3 - 5 times per day as tolerated
  Other Names: Allergy Research Group is supplying the placebo tablets.
  Arms: 2

SUMMARY:
Participants will be diagnosed with localized prostate or breast cancer and be scheduled to undergo external beam radiation therapy. Participants will either receive a placebo or organic germanium to be taken 5 times a day starting the day of their first radiation and continuing through the 1 month follow-up visit. Weekly Quality of life forms will be completed through the one month follow up visit and then at the 3 month follow up visit. Labs will be done prior to the start of treatment, at the end of treatment and at the one and three month follow-up visits.

DETAILED DESCRIPTION:
With the increasing public use of complementary medicines, most researchers agree that there is a compelling need to study the safety and efficacy of these agents in humans by means of appropriately designed double-blind, placebo controlled clinical trials. With fatigue affecting 96% of the cancer patient population and little more than life style alterations offered as an intervention, the need to evaluate putative and innovative approaches for fatigue is a high priority. The NIH released a "State of the Science" statement in 2002 which concluded that fatigue is a serious cause of morbidity, being the most prevalent symptom experienced by cancer patients. This expert panel also concluded that the major barrier to effective management of fatigue includes a lack of awareness of this fact, the lack of knowledge of the causes of fatigue, and the lack of proven methods to treat fatigue. Presently, clinical trials evaluating intervention for cancer fatigue are lacking.

Organic germanium literature states that it may be an effective agent for combating fatigue with virtually no toxicities. Since virtually all cancer patients receiving radiation therapy experience fatigue, the use of this drug should be evaluated as an intervention for non-anemic fatigue in breast and prostate cancer patients undergoing a definitive course of radiation therapy. We intend to test whether organic germanium is able to reduce the fatigue experienced by patients undergoing radiation therapy and if this reduction in fatigue correlates to an improvement in quality of life for these patients. Changes in the patients' mood will also be evaluated. We will also collect information on the toxicity profile of Organic germanium and try to determine when the peak fatigue time occurs and possibly when they recover. This information will be utilized to see if a larger study is warranted.

2.0 OBJECTIVES 2.1 Primary: To determine if Organic germanium is effective in decreasing severity of fatigue in patients undergoing definitive radiation therapy for prostate or breast cancer at the one month follow-up visit.

2.2 Secondary 2.2.1 To compare changes in patients' moods between Organic germanium versus placebo at the one month follow-up visit 2.2.2 To compare the duration of fatigue between organic germanium and placebo 2.2.3 To further evaluate the toxicity profile of organic germanium using the CTCAE version 3 scale.

2.2.4 To determine the Peak time of fatigue in patients receiving external beam radiotherapy or high dose rate brachytherapy for breast or prostate cancer.

2.2.5 To determine the tolerability of 5 tablets per day as the dosing schema. 2.2.6 To determine when the patients recover from their radiation induced fatigue

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed diagnosis of breast (females only) or prostate cancer
2. Zubrod performance status of 0-1.
3. Patients must be ≥ 18 years of age.
4. Scheduled to undergo definitive radiation therapy (either brachytherapy or external beam)
5. Patients may have received or be receiving hormonal therapy. Prior chemotherapy is allowed as long as the patient has recovered from any toxicity. Planned future chemotherapy is also allowed after the one month evaluation.
6. Hgb ≥ 10 g/dl, BUN < 25 mg and creatinine < 1.5 mg
7. Patient must be able to comply with treatment regimen.
8. Patient must complete the pre-treatment quality of life questionnaires.
9. Women of childbearing potential must have a pre-treatment pregnancy test; women of childbearing potential and men able to father children must use non-hormonal-based birth control while on study.
10. Patients must sign study-specific informed consent prior to study entry.

Exclusion Criteria:

1. Known allergies or reactions to Organic germanium
2. Prior irradiation other than basal cell cancer of skin
3. Current or past history of metastasis
4. Current history of uncontrolled hypertension, insulin dependent or uncontrolled diabetes, cardiovascular disease unless controlled and stable for 6 months or more, bleeding disorders, or autoimmune disorders such as fibromyalgia, chronic fatigue syndrome or lupus
5. Current use of corticosteroids or erythropoietin
6. Patients currently taking Organic germanium, or who have taken Organic germanium within the past three months
7. Pregnant or lactating women, as treatment involves unforeseeable risks to the participant and to the embryo or fetus
8. Patients who are unable to complete quality of life questionnaires
9. Male breast cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2005-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine if Organic germanium is effective in decreasing severity of fatigue in patients undergoing definitive radiation therapy for prostate or breast cancer at the one month follow-up visit. | One month pst treatment

SECONDARY OUTCOMES:
To compare changes in patients' moods between Organic germanium versus placebo at the one month follow-up visit | One month follow up
To compare the duration of fatigue between organic germanium and placebo | One month follow up
To further evaluate the toxicity profile of organic germanium using the CTCAE version 3 scale. | one month follow up
To determine the Peak time of fatigue in patients receiving external beam radiotherapy or high dose rate brachytherapy for breast or prostate cancer. | one month follow up
To determine when the patients recover from their radiation induced fatigue | 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Emily Grade, MD, Principal Investigator — Arizona Oncology Services
Locations (1):
- Arizona Oncology Services, Phoenix, Arizona, United States

REFERENCES:
- See also: Related Info — http://www.azoncology.com/internet/AOSFoundationClinicalTrials/ClinicalTrials/BreastCancerStudies/tabid/64/Default.aspx
- See also: Related Info — http://www.azoncology.com/internet/ResearchClinicalTrials/ClinicalTrials/GenitourinaryStudies/tabid/66/Default.aspx